CLINICAL TRIAL: NCT05664789
Title: Targeting the Neurobiology of Restricted and Repetitive Behaviors in Children With Autism Using N-acetylcysteine: A Randomized, Controlled Trial
Brief Title: Targeting the Neurobiology of RRB in Autism Using N-acetylcysteine: Trial
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Patrick Hegarty, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-68353; 4R00HD101702-03 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Magnetic resonance imaging; N-acetyl cysteine; Restricted and repetitive behaviors; Electroencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled trial 2 arms, N-acetylcysteine and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo compound will match the active N-acetylcysteine in appearance, odor, taste, and packaging.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- N-acetylcysteine (Active Comparator): 12 week administration of active study compound
  Interventions: Drug: N acetyl cysteine
- Placebo (Placebo Comparator): 12 week administration of matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N acetyl cysteine — N-acetylcysteine (NAC) is an over-the-counter dietary supplement that is relatively well tolerated and exhibits minimal side effects, even at high dosages. N
  Arms: N-acetylcysteine
Drug: Placebo — matched placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to target the neurobiology of restricted and repetitive behaviors in children with autism spectrum disorder using N-acetylcysteine (NAC), a well-tolerated nutritional supplement that has shown promise for reducing symptom severity in recent small-scale trials. The findings from this research will shed light on the mechanisms of action underlying the clinical benefits of NAC and the effects of NAC on altering restricted and repetitive behavior symptom severity in children with autism spectrum disorder. This is a 12-week double-blind, randomized, placebo-controlled trial of NAC.

ELIGIBILITY:
Inclusion Criteria:

* children between 3 years and 12 years 11 months
* diagnosis of autism spectrum disorder confirmed with the Autism Diagnostic Interview- Revised and the Autism Diagnostic Observation Schedule-2, Brief Observation of Symptoms of Autism, or Childhood Autism Rating Scale
* at least moderate severity of restricted and repetitive behaviors defined by a Children's Yale-Brown Obsessive Compulsive Scale for Autism Spectrum Disorder score ≥ 11
* physical development indicative of prepubescence as defined by criteria for Tanner Stage 1
* if home address is within 300 miles of the primary study site, participants must pass MR safety screening (e.g., no metal in the body) and attempt baseline neuroimaging (MRI or EEG), otherwise baseline neuroimaging is not required for participation
* have stable medication regimens (≥ 30 days) and psychosocial treatments (≥ 60 days) prior to randomization with no anticipated changes during the trial

Exclusion Criteria:

* presence of known genetic abnormalities associated with ASD (e.g. Fragile X)
* current or life-time diagnosis of severe psychiatric disorder (e.g., schizophrenia)
* presence of significant medical problems
* the inability of at least one caregiver to speak and read English to a sufficient level
* participants taking glutathione agents/prodrugs
* history of any adverse effects to glutathione agents/prodrugs
* the inability to drink a sample study compound dissolved in liquid

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Children's Yale Brown-Obsessive Compulsive Scale for Autism Spectrum Disorder (CYBOCS-ASD) at 12 weeks | Screening and week 12
  Severity of restricted and repetitive behaviors, higher scores indicate more severe behaviors
Change in Glutamatergic neurometabolites at 12 weeks | Baseline and week 12
  Glu and Glx measured by magnetic resonance imaging

SECONDARY OUTCOMES:
Change in Restricted and Repetitive Behavior Scale Revised (RBS-R) at 12 weeks | Baseline and week 12
  Severity of restricted and repetitive behaviors, higher scores indicate more severe behaviors
Change in Gamma band activity at 12 weeks | Baseline and week 12
  Electrical activity between 30-48 Hz measured by electroencephalography

CONTACTS AND LOCATIONS:
Overall Officials: John Hegarty, PhD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be shared with the National Database for Autism Research (NDAR)
Time Frame: The data will be shared on January 15th and July 15th each year
Access Criteria: Researchers with access to the National Database for Autism Research (NDAR) will be able to obtain the submitted data
URL: http://nda.nih.gov